CLINICAL TRIAL: NCT07006246
Title: Utilizing Private Pharmacies to Initiate High Risk Young Women and Men on Pre-exposure Prophylaxis (PrEP) in South Africa
Brief Title: Utilizing Private Pharmacies to Initiate High-risk Young Individuals on PrEP in South Africa
Acronym: PPREPP-SA
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Professor Francois Venter (Other)
Collaborators: Bill and Melinda Gates Foundation (Other)
Responsible Party: Sponsor-Investigator, Professor Francois Venter, Executive Director: Ezintsha, University of Witwatersrand, South Africa
Organization: University of Witwatersrand, South Africa (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: EZ-FV-032
Record Dates: First submitted 2025-03-25; First posted 2025-06-05 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-05

CONDITIONS: HIV Infection
Keywords: tenofovir disoproxil fumarate/emtricitabine (TDF/FTC); pre-exposure prophylaxis (PrEP); Private Pharmacies; Implementation study
MeSH Terms: conditions — HIV Infections | interventions — Tenofovir; Lamivudine; Emtricitabine; Racivir

STUDY DESIGN:
Intervention Model Description: This is a two-stage (formative and implementation) implementation study. We will employ a mixed-method approach-specifically, a divergent parallel design. We will use the EPIS framework (Exploration, Preparation, Implementation, and Sustainability) as an overarching implementation structure to Formalize stakeholder partnerships and tailor the proposed service delivery models (intervention package) for the implementation context.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Tenofovir disoproxil fumarate + lamivudine/emtricitabine (TDF+3TC /FTC) (Other): Dosage Formulation: 300 mg / 200 mg (300mg) fixed dose combination tablet Route of Administration: Oral Dosing Instructions: 1 tablet (300/200/ TDF/FTC) daily or (300/300/TDF/3TC) daily
  Interventions: Drug: Tenofovir disoproxil fumarate + lamivudine/emtricitabine (TDF+3TC /FTC)

INTERVENTIONS:
Drug: Tenofovir disoproxil fumarate + lamivudine/emtricitabine (TDF+3TC /FTC) — Tenofovir disoproxil fumarate + emtricitabine/ lamivudine Dosage Formulation: 300 mg / 200 mg (300mg) fixed dose combination tablet Route of Administration: Oral Dosing Instructions: 1 tablet (300/200/ TDF/FTC) daily or (300/300/TDF/3TC) daily

SUMMARY:
This is a funded implementation study designed to evaluate the efficacy of recruiting and retaining high-risk individuals on pre-exposure prophylaxis (PrEP) within multiple private pharmacies (and online platforms in South Africa)

DETAILED DESCRIPTION:
This is a two-stage (formative and implementation) study. It will employ a mixed-method approach-specifically, a divergent parallel design. The study will use the EPIS framework (Exploration, Preparation, Implementation, and Sustainability) as an overarching implementation structure to Formalise stakeholder partnerships and tailor the proposed service delivery models (intervention package) for the implementation context.

The study chose EPIS as it considers the multilevel nature of healthcare, organizations within systems, and patient needs. Using the capability, opportunity, and motivation for behaviour (COM-B) change model, the study will assess the readiness of pharmacists, pharmacy nurses, and pharmacy clinics to adopt and implement the service delivery models. The study will use participatory human-centred stakeholder engagement to inform appropriateness, acceptability, and feasibility of the service delivery models, priorities for tailoring, and responsibilities for implementation.

As a multi-centre pharmacy-initiated implementation study, the project is designed to assess the feasibility and acceptability of in-pharmacy oral PrEP initiation, and oral PrEP initiation utilizing a virtual model and in-pharmacy administration. Additionally, this study will provide information about tolerability, safety, and preferences on accessing prophylactic HIV services. In the formative phase, cross-sectional data collection will take place, while during the implementation stage, young women and men will be screened and recruited to the study across sites in Gauteng and the Western Cape and will be followed over 13 months (prospective, longitudinal).

ELIGIBILITY:
Inclusion Criteria:

* Adult male or female (≥18 and ≤ 35 years old)
* HIV negative at the time of study enrolment (as determined by a rapid blood test for HIV 1,2)
* Absence of symptoms of acute HIV infection*
* Body weight ≥ 35 kg
* Creatinine clearance ≥ 50 mL/min
* Willingness to take PrEP as prescribed and to comply with study procedures.
* Willingness to be followed up throughout the duration of the study.

Exclusion Criteria:

* Confirmed HIV positive by routine antibody testing
* Presence of symptoms of acute HIV infection*
* Creatinine clearance (eGFR) of:

  * Less than 50 mL/min/1.73m2 for adults
  * For pregnant women: serum creatinine (sCr) greater than 85 µmol/L
* Known hypersensitivity to or specific contraindications to the use of TDF or FTC/3TC
* Self-reported presence or history of liver cirrhosis (Child-Pugh Class B or greater), with or without viral hepatitis co-infection
* Any surgical or medical condition which may significantly alter the absorption, distribution, metabolism, or excretion of drugs, or which may jeopardize the safety of the participant. This will be an investigator-led determination based on the medical history of the participant. This includes, but is not limited to:

  • Severe hepatic impairment or history of liver cirrhosis with or without viral hepatitis co-infection.
* Participant is judged by the Investigator to be at significant risk of failing to comply with the provisions of the protocol as to cause harm to self or seriously interfere with the validity of the study results.
* Inability or unwillingness to be followed up for the study period
* Pregnant and lactating women

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1900 (Estimated)
Dates: Start 2023-05-19 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Number of pharmacies providing Prep services over 13 months | 13 Months
  Acceptability of pharmacy-delivered PrEP services will be determined by qualitative and quantitative assessment using piloted and validated semi-structured questionnaires for acceptability.
Number of participants accessing PrEP online services over 13 months | 13 Months
  Acceptability of online-delivered PrEP services will be determined by qualitative and quantitative assessment using piloted and validated semi-structured questionnaires for acceptability.

SECONDARY OUTCOMES:
To describe provider experiences and perceptions of pharmacy and online-delivered PrEP | 13 Months
  Provider Perspectives on service delivery using semi-structured interviews using REAIM
To describe user experiences and perceptions of pharmacy and online-delivered PrEP | 13 Months
  User perspectives on service delivery using semi-structured interviews using REAIM

CONTACTS AND LOCATIONS:
Overall Officials: Fanscois Venter, PhD in Medicine, Principal Investigator — Ezintsha, a subdivision of Wits Health Consortium
Locations (1):
- Ezintsha, a division of Wits Health Consortium, Johannesburg, Gauteng, South Africa

IPD SHARING:
Plan to Share IPD: Yes
After deidentification, the data will be shared with the study participants of the trial.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: After the study results are published
Access Criteria: Anyone who needs to access the data